CLINICAL TRIAL: NCT03378674
Title: Effect of Different Doses of Remifentanil on Stress Response During Laparoscopic Cholecystectomy
Brief Title: Remifentanil and Stress Hormones Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Germano De Cosmo, professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CUSacredHeart
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Stress Response
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): remifentanil infusion of 0,15 mcg/Kg/min
  Interventions: Drug: Remifentanil Injectable Product
- Group B (Active Comparator): remifentanil infusion of 0,3 mcg/Kg/min
  Interventions: Drug: Remifentanil Injectable Product

INTERVENTIONS:
Drug: Remifentanil Injectable Product — remifentanil: 0,15 mcg/kg/min

SUMMARY:
Perioperative adequate analgesia reduces neuroendocrine stress response and postoperative complications. Because opioids are the most effective parenteral drugs to control pain and stress response, in this prospective randomized double-blinded controlled study we supposed that higher dose of remifentanil may reduce stress marker variations compared to lower dose in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Fifty Caucasian patients, aged 20-70 years, with American Society of Anesthesiologist physical status I-II, undergoing laparoscopic cholecystectomy were enrolled. Exclusion criteria were: patient refusal, thyroid disorders, diabetes mellitus, BMI > 30, use of corticosteroids, benzodiazepines or antipsychotics drugs. No patient received premedication. Before entering the operating room, venous access was established (18 G in the antecubital vein) where the first blood sample (Time 0) was collected to measure adrenocorticotropic hormone (ACTH), Cortisol, Growth hormone (GH) and prolactin (PRL) levels. Then a second venous access was established (18 G on the other arm) to start a fluid infusion (normal saline to replace half of the water deficit from preoperative fasting followed by a maintenance infusion of 2 ml/kg/h). Heart Rate (HR), Non Invasive Blood Pressure (NIBP), Bispectral Index (BIS), End-tidal CO2 (EtCO2) were recorded every 5 minutes. Patients were randomly assigned to receive two different dosages of remifentanil: 0,15 mcg/kg/min (group A) and 0,30 mcg/kg/min (group B) for the induction and the maintenance of anesthesia, using a computer generated randomization table (Table I). Anesthesia was induced with propofol 2 mg/kg, cisatracurium 0,15 mg/kg and remifentanil infusion of 0,15 mcg/Kg/min (Group A) or 0,3 mcg/Kg/min (Group B) was started. Anesthesia was maintained with desflurane at a variable concentration in order to maintain the BIS between 40 and 60. The second blood sample was collected at the trocar insertion (Time 1), and the third sample one hour after the end of the surgery (Time 2). Postoperative analgesia was standardized using intravenous acetaminophen 1 g and morphine 0,1 mg/kg 30 minutes before the end of the surgery. Rescue analgesia in Recovery Room was provided by intravenous tramadol 1 mg/Kg.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist physical status I-II
* Undergoing laparoscopic cholecystectomy

Exclusion Criteria:

* patient refusal,
* thyroid disorders,
* diabetes mellitus,
* BMI > 30,
* use of corticosteroids, benzodiazepines or antipsychotics drugs

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
ACTH levels changes | changes between basal, incision,one hour after surgery
Cortisol levels changes | changes between basal, incision,one hour after surgery
Growth hormone levels changes | changes between basal, incision,one hour after surgery
prolactin levels changes | changes between basal, incision,one hour after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Flaminio Sessa, MD, Principal Investigator — Catholic University Rome
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy

REFERENCES:
- [Background] Jakeways MS, Mitchell V, Hashim IA, Chadwick SJ, Shenkin A, Green CJ, Carli F. Metabolic and inflammatory responses after open or laparoscopic cholecystectomy. Br J Surg. 1994 Jan;81(1):127-31. doi: 10.1002/bjs.1800810146. PMID 8313088
- [Background] Marana E, Scambia G, Maussier ML, Parpaglioni R, Ferrandina G, Meo F, Sciarra M, Marana R. Neuroendocrine stress response in patients undergoing benign ovarian cyst surgery by laparoscopy, minilaparotomy, and laparotomy. J Am Assoc Gynecol Laparosc. 2003 May;10(2):159-65. doi: 10.1016/s1074-3804(05)60291-5. PMID 12732764
- [Background] Adas G, Kemik A, Adas M, Koc B, Gurbuz E, Akcakaya A, Karahan S. Metabolic and inflammatory responses after ERCP. Int J Biomed Sci. 2013 Dec;9(4):237-42. PMID 24711760
- [Background] Desborough JP. The stress response to trauma and surgery. Br J Anaesth. 2000 Jul;85(1):109-17. doi: 10.1093/bja/85.1.109. No abstract available. PMID 10927999